CLINICAL TRIAL: NCT00002110
Title: A Phase II/III Study of Cysteamine (Mercaptoethylamine) and Zidovudine for the Treatment of HIV Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mylan Laboratories (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: Double | Purpose: Treatment
Other Study IDs: 211A; CYST-9304
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1995-10

CONDITIONS: HIV Infections
Keywords: Drug Therapy, Combination; AIDS-Related Complex; Zidovudine; Cysteamine
MeSH Terms: conditions — HIV Infections; AIDS-Related Complex | interventions — Cysteamine; Zidovudine

INTERVENTIONS:
Drug: Cysteamine
Drug: Zidovudine

SUMMARY:
To determine the safety and tolerance of low-dose versus high-dose cysteamine administered concurrently with zidovudine (AZT). To determine the pharmacokinetics and effects on immune function and viral load in patients receiving these drug regimens.

DETAILED DESCRIPTION:
Patients receive high or low doses of cysteamine plus AZT or placebo plus AZT. The target dose of cysteamine is determined by titration of the dose over a 6-week period, after which the patient receives 24 additional weeks of treatment. An initial cohort of 36 patients will be enrolled in a 10-week pilot phase. Accrual will be temporarily suspended while data from the pilot phase is assessed.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Chemoprophylaxis for Pneumocystis carinii pneumonia, candidiasis, Mycobacterium tuberculosis, and herpes as prescribed by the investigator.
* Recombinant erythropoietin and G-CSF if clinically indicated.

Patients must have:

* Documented HIV infection.
* CD4 count 300 - 500 cells/mm3.
* Prior AZT therapy for at least 3 months but less than 12 months prior to study entry.
* No past or current AIDS-defining opportunistic infection.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Kaposi's sarcoma requiring systemic therapy.
* Active malignancy other than basal cell carcinoma or in situ cervical carcinoma.

Concurrent Medication:

Excluded:

* Antiretroviral therapy other than AZT.
* Immunosuppressive drugs.
* Investigational HIV drugs/therapies other than study drug.
* Interferon.
* Steroids.
* Hematopoietins.
* Cytotoxic chemotherapy including Adriamycin, bleomycin, and vincristine.

Concurrent Treatment:

Excluded:

* Radiation therapy.

Patients with the following prior condition are excluded:

History of treatment-limiting intolerance to 500-600 mg AZT daily as manifested by the same recurrent grade 3 toxicity or any prior grade 4 toxicity.

Prior Medication:

Excluded:

* Prior antiretroviral therapy other than AZT.

Required:

* AZT for at least 3 months but no more than 12 months prior to study entry.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Infectious Disease Research Institute Inc, Tampa, Florida
  - Tulane Univ Med School, New Orleans, Louisiana
  - SUNY / Health Sciences Ctr at Stony Brook, Stony Brook, New York
  - Bowman Gray School of Medicine / North Carolina Baptist Hosp, Winston-Salem, North Carolina
  - Independent Research Nurses Inc, Cranston, Rhode Island
  - Univ of Texas Southwestern Med Ctr of Dallas, Dallas, Texas